CLINICAL TRIAL: NCT05580926
Title: Evaluation of the Efficacy of the Watch Your Weight During Holidays Program for the Prevention of Body Weight Gain in Mexican Adults: Two-arm Randomized Controlled Trial With Parallel Groups.
Brief Title: Evaluation of the Efficacy of the Watch Your Weight During Holidays Program for the Prevention of Body Weight Gain in Mexican Adults.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rolando Giovanni Díaz Zavala (Other)
Responsible Party: Sponsor-Investigator, Rolando Giovanni Díaz Zavala, Research Professor, Universidad de Sonora
Organization: Universidad de Sonora (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USO313008171
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Obesity; Weight Gain; Overweight
Keywords: Holiday Season; Prevention
MeSH Terms: conditions — Obesity; Weight Gain; Overweight | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors of the variables of interest will be blinded to the allocation group. The person responsible for randomization will be external, not involved in recruitment, study measurements and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Watch your Weight During Holidays Program (Experimental)
  Interventions: Behavioral: Watch your Weight During Holidays
- Control group (minimal intervention) (Placebo Comparator)
  Interventions: Other: Control Group (minimal intervention)

INTERVENTIONS:
Behavioral: Watch your Weight During Holidays — Participants in this group will have an individual face-to-face session (with a maximum duration of half an hour) and a face-to-face group session. This intervention will include strategies for self-monitoring (body weight, diet and physical activity), information on healthy lifestyles, as well as information about the energy contained in local festive foods and their equivalent in minutes of physical activity or steps per day.
  Participants will be asked to weight themselves at least twice a week, as a form of self-monitoring of weight, from the start of the intervention. They will have access to weekly forms with boxes, where they can fill in the data obtained for each day of weight self-monitoring, energy intake restriction report and minutes of physical activity performed.
  Arms: Watch your Weight During Holidays Program
Other: Control Group (minimal intervention) — Participants in this group will receive a printed information, as well as a PDF file, brochure during a face-to-face session at the beginning of the 8-week period. This information will be about having a healthy eating based on the norm for health promotion and education for healthy eating in Mexico (NOM-043-SSA2-2012).
  Arms: Control group (minimal intervention)

SUMMARY:
Obesity is the main risk factor for the development of chronic-degenerative diseases in Mexico. Due to the difficulty of treating obesity, prevention is urgently needed. The holidays are the festive period with the greatest impact on adult body weight. Evidence from observational studies has shown that more than 50% of the annual weight is gained during this period. However, few preventive interventions have been carried out worldwide. The present work will evaluate the efficacy of the Watch your Weight During Holidays Program on the prevention of weight gain during 8 weeks in comparison with the control group in Mexican adults. The study will be a randomized clinical trial. It will have two intervention groups: 1) Watch your Weight During Holidays Program and 2) Control Group (minimal intervention). Weight, height, body mass index, waist circumference, kilograms of body fat, fat mass index, cm2 of abdominal fat, blood pressure and perception of health-related quality of life will be measured in 64 volunteers, at the beginning and after 8 weeks of participating in Watch your Weight During Holidays Program. For comparisons between groups, Student's t-tests or Mann-Whitney's U-tests will be performed, according to the type of sample distribution. The primary variable of the study will be the change in body weight. The secondary variables will be the change in body mass index, waist circumference, kilograms of fat mass, fat mass index, cm2 of abdominal fat, blood pressure and aspects of perception of quality of life related to health.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 and ≤60 years of age).
* Residents of the city of Hermosillo, Sonora.
* BMI ≥ 23 and ≤ 40.
* Availability of time to participate in the study, including initial and final measurements.
* Have a device with access to WhatsApp
* Accept not to carry out any other intervention outside of the one assigned in the study during the 8 weeks of the intervention.

Exclusion Criteria:

* Have medical conditions due to previous diagnosis, which require the prescription of treatments that affect weight, such as diabetes and thyroid diseases.

Other exclusion criteria will be liver failure, cancer under treatment or at an advanced stage, a history of COVID-19 that has required hospitalization, supplemental oxygen or left sequelae that contraindicate the intervention; psychiatric conditions, eating disorders, etc.

* Use of drugs or substances with an effect on weight, for example, metformin, orlistat, corticosteroids, etc.
* Use of addictive substances such as drugs of abuse
* Previous bariatric surgery.
* Being a participant in another intervention or treatment for the management of obesity.
* Weight loss > 5% of total body weight in the last 4 months.
* Having plans to become pregnant within the study period, currently pregnant or breastfeeding.
* Another family member has agreed to participate in the study.
* Illiteracy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-10-11 (Estimated); Primary Completion 2023-01-13 (Estimated); Study Completion 2023-01-13 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight | Baseline to 8 weeks

SECONDARY OUTCOMES:
Changes in body mass index | Baseline to 8 weeks
Changes in waist circumference | Baseline to 8 weeks
Changes in kilograms of body fat | Baseline to 8 weeks
Changes in body fat index | Baseline to 8 weeks
Changes in cm2 of abdominal fat | Baseline to 8 weeks
Changes in systolic blood pressure | Baseline to 8 weeks
Changes in diastolic blood pressure | Baseline to 8 weeks
Changes in perception of health related quality of life | Baseline to 8 weeks
  The SF-36 Health Survey evaluates aspects of the quality of life in adult populations (over 16 years of age). The result of its application is the generation of eight concepts or scales of health, result of the average of the sum of the questions contained in the questionnaire for each concept. These concepts are: physical function, physical role, corporal pain, general health, vitality, social function, emotional role and mental health. The SF-36 is a self-applied instrument and contains 36 questions. For each scale, the answers to each question are coded and recoded (10 questions), and the results are interpreted on a scale of 0 to 100, lower results indicate poorer health and greater result better health.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Promoción de Salud Nutricional (CPSN), Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: Undecided